CLINICAL TRIAL: NCT06725862
Title: Comparison of the Effects of Caudal Block and Retrolaminar Block on Analgesic Consumption in Postoperative Pain Management for Pediatric Undescended Testis Surgeries
Brief Title: Caudal Block vs Retrolaminar Block on Analgesic Consumption in Undescended Testis Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Engin Ihsan Turan, anesthesiology and reanimation specialist, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: caudal vs retrolaminar
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrolaminar block group (Experimental): Pediatric patients in this group will receive a retrolaminar block (RLB) using 0.25% bupivacaine (0.1 mL/kg) injected into the retrolaminar space at the L4 vertebral level under ultrasound guidance after general anesthesia induction.
  Interventions: Procedure: Retrolaminar Block (RLB)
- Caudal Block (CB) Group (Active Comparator): Pediatric patients in this group will receive a caudal block (CB) using 0.125% bupivacaine (1 mL/kg, maximum 20 mL) injected into the sacral canal under ultrasound guidance after general anesthesia induction.
  Interventions: Procedure: Caudal Block (CB)

INTERVENTIONS:
Procedure: Retrolaminar Block (RLB) — This intervention involves administering 0.25% bupivacaine (0.1 mL/kg) into the retrolaminar space at the L4 vertebral level using a 22-G insulated needle under ultrasound guidance in pediatric patients after induction of general anesthesia.
  Arms: Retrolaminar block group
Procedure: Caudal Block (CB) — This intervention involves administering 0.125% bupivacaine (1 mL/kg, maximum 20 mL) into the sacral canal using a 22-G insulated needle under ultrasound guidance in pediatric patients after induction of general anesthesia.
  Arms: Caudal Block (CB) Group

SUMMARY:
This study compares the postoperative analgesic effectiveness of Caudal Block (CB) and Retrolaminar Block (RLB) in pediatric patients undergoing undescended testis surgeries. Both techniques aim to manage pain effectively and reduce reliance on systemic analgesics, improving recovery and minimizing complications.

The double-blind, randomized controlled trial will include 1-7-year-old ASA I-II patients at two hospitals. Patients with specific contraindications (e.g., spinal anomalies, allergies, or infections) will be excluded. Randomization divides participants into two groups (CB and RLB), with pain assessments performed using the FLACC pain scale by a blinded nurse.

Procedures:

CB: 0.125% bupivacaine (1 mL/kg, max 20 mL) injected into the sacral canal under ultrasound guidance.

RLB: 0.25% bupivacaine (0.1 mL/kg) injected into the retrolaminar space at the L4 level under ultrasound guidance.

Postoperative pain will be evaluated at various intervals (30 minutes to 24 hours). Intravenous paracetamol or tramadol will be administered based on pain scores.

The study aims to compare pain scores, time to first analgesic requirement, and postoperative complications, contributing valuable data on these two regional anesthesia techniques in pediatric surgery.

DETAILED DESCRIPTION:
Pediatric lower abdominal surgeries, especially undescended testis surgeries, are procedures that can cause significant pain in the postoperative period. Effective pain management in such surgeries is crucial to accelerate recovery in children and reduce complications associated with analgesic medications. Among the most commonly used regional anesthesia techniques for pediatric lower abdominal surgeries is the caudal block, which has provided effective pain management for many years. However, in recent years, ultrasound-guided trunkal nerve blocks have gained popularity due to their targeted and prolonged analgesic effects. One such block, the retrolaminar block (RLB), is a relatively new technique applied around the spinal laminae with local anesthetics and has been increasingly utilized in pediatric surgeries.

While the caudal block is widely used in lower abdominal surgeries, ensuring proper distribution of the anesthetic agent and monitoring for potential side effects during the procedure is necessary. In contrast, the retrolaminar block, performed reliably under ultrasound guidance, is suggested to provide longer-lasting analgesia compared to the caudal block. The RLB allows for broader spread of the local anesthetic in the paraspinal region, potentially affecting both lower and upper areas. However, studies comparing the postoperative analgesic effects of RLB and caudal block in pediatric patients are quite limited in the literature.

This study aims to compare the postoperative analgesic effectiveness of caudal block and retrolaminar block in pediatric patients undergoing undescended testis surgeries. The study evaluates differences between these two regional anesthesia techniques in terms of postoperative pain scores, time to first analgesic requirement, and postoperative complications. The limited data available on these block methods in the literature highlight the potential scientific contribution of this study.

This double-blind, randomized controlled trial will be conducted at Prof. Dr. Cemil Taşçıoğlu City Hospital and Zincirlikuyu Medicana Hospitals. Following clinical ethics committee approval, the study will include pediatric patients aged 1 to 7 years who are classified as ASA I-II and scheduled for unilateral undescended testis surgeries.

Patients under 1 year or over 7 years, those with neurological deficits, bleeding disorders, a history of allergies to local anesthetics, signs of redness or infection at the injection site during physical examination, congenital spinal anomalies, mental retardation, psychiatric disorders, liver or kidney disease, and those who do not consent to participate will be excluded from the study.

Randomization and blinding Randomization will be performed using a computer-generated randomization table, dividing patients into two groups: Retrolaminar Block (RLB) and Caudal Block (CB). Pain evaluation will be conducted using the FLACC pain scale, assessed by a blinded nurse. The anesthesiologist will be blinded to data collection related to analgesic requirements and postoperative complications. Transparent sterile drapes will be applied to all injection sites to blind the anesthesiologist to postoperative outcomes.

General anesthesia procedure All patients will receive 0.5 mg/kg oral midazolam as premedication. Following standard monitoring in the operating room, general anesthesia will be induced with 2 mg/kg intravenous propofol and 0.5 μg/kg fentanyl. After loss of the eyelash reflex, a laryngeal mask airway suitable for the patient's age and weight will be inserted without using muscle relaxants, and the patient will be connected to the anesthesia machine. Anesthesia will be maintained with 2% sevoflurane in a 50% air-oxygen mixture. Demographic data (age, weight, duration of surgery) and complications will be recorded.

Regional anesthesia procedure Blocks will be performed in the left lateral decubitus position under ultrasound guidance by a single experienced operator after induction of general anesthesia and securing the airway. A 22-G insulated 50-mm sonographic needle will be used for all injections. Ultrasound guidance will be performed using a linear probe (6.5-18 MHz) in nerve imaging mode.

Caudal Block (CB) procedure The surgical area will be sterilized with povidone-iodine. The sacral hiatus will be visualized using the out-of-plane transverse imaging technique, and 0.125% bupivacaine at a dose of 1 mL/kg (maximum 20 mL) will be injected into the sacral canal.

Retrolaminar Block (RLB) procedure Patients will be positioned in the left lateral decubitus position. Using a paramedian sagittal approach at the L4 vertebral level, the transverse process of L4 will be located with the ultrasound probe. A needle will then be advanced into the retrolaminar space between the L4 lamina and paraspinal muscles, and 0.25% bupivacaine at a dose of 0.1 mL/kg will be injected.

Caudal block has long been used as a method of pain relief in pediatric anesthesia, significantly improving postoperative comfort, relieving pain, and reducing side effects such as nausea and vomiting. Similarly, retrolaminar block, which is among the routine practices in our hospital, enhances postoperative comfort by better controlling pain. This technique provides safe and effective analgesia by targeting nerves through injections into the lamina region of the spine while minimizing spread to surrounding tissues. The efficacy and reliability of retrolaminar block support its preference in postoperative pain management.

Postoperative follow-up and pain evaluation Pain will be assessed using the FLACC pain scale at 30 minutes, and at 1, 2, 4, 6, 12, and 24 hours. Patients with scores of 2-4 will receive intravenous paracetamol, and those with scores above 4 will be given intravenous tramadol. The timing and amount of analgesic use will be recorded.

ELIGIBILITY:
Inclusion Criteria:

Pediatric patients aged 1-7 years. ASA (American Society of Anesthesiologists) physical status I or II. Scheduled for unilateral undescended testis surgery. Parental/guardian consent provided for study participation.

Exclusion Criteria:

Age under 1 year or over 7 years. Neurological deficits. Coagulopathy or bleeding disorders. History of allergy to local anesthetics. Signs of redness, infection, or other abnormalities at the injection site. Congenital spinal anomalies. Intellectual disability or psychiatric disorders. Hepatic or renal impairment. Refusal to participate in the study by parents or guardians.

Ages: 1 Year to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-16 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Scores | Up to 24 hours postoperatively.
  Assessment of postoperative pain scores using the FLACC scale (Face, Legs, Activity, Cry, Consolability) at predefined intervals (30 minutes, 1, 2, 4, 6, 12, and 24 hours postoperatively). Scores range from 0 to 10, with higher scores indicating greater pain intensity.

SECONDARY OUTCOMES:
Time to First Analgesic Requirement | Up to 24 hours postoperatively.
  The time elapsed from the completion of the surgical procedure to the first administration of rescue analgesia (IV paracetamol or tramadol) based on FLACC scores.
Total Analgesic Consumption | Up to 24 hours postoperatively.
  The cumulative amount of analgesic medications (paracetamol and/or tramadol) administered within the first 24 hours postoperatively.
Incidence of Postoperative Complications | Up to 24 hours postoperatively.
  The occurrence of complications such as nausea, vomiting, or urinary retention associated with the analgesic techniques used.

CONTACTS AND LOCATIONS:
Overall Officials: Engin ihsan Turan, Principal Investigator — Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital, Istanbul
  - Zincirlikuyu Medicana Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided